CLINICAL TRIAL: NCT00962793
Title: Diagnosis of Latent Tuberculosis(TB) Infection in Health Care Workers Using TST and Whole Blood Interferon-γ Assay
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Other Study IDs: 4-2009-0187
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2009-08-20 (Estimated); Status verified 2009-08

CONDITIONS: Tuberculosis
Keywords: latent tuberculosis prevalence of health care workers
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The investigators think that the health care workers who contact frequently with active tuberculosis patients have more increased prevalence of LTBI compared with those who don't.

ELIGIBILITY:
Inclusion Criteria:

* health care workers

Exclusion Criteria:

* active pulmonary tuberculosis
* previous Tuberculosis history
* below 20 years old
* history of hypersensitivity about PPD
* pregnant

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: latent tuberculosis prevalence of health care workers
Sampling Method: Probability Sample